CLINICAL TRIAL: NCT00827541
Title: A Phase IV Pharmacovigilance, Post-Authorization Clinical Trial To Evaluate And Assess The Safety Of Tigecycline In The Approved Indications In The Usual Health Care Setting
Brief Title: Post-Authorization Study Evaluating Safety Of Tigecycline
Acronym: HORUS
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1811048; 3074A1-4401
Record Dates: First submitted 2009-01-20; First posted 2009-01-22 (Estimated); Results first posted 2012-02-01 (Estimated); Last update posted 2012-02-01 (Estimated); Status verified 2011-12

CONDITIONS: Intra-Abdominal Infections; Skin Disease, Infectious; Soft Tissues Infections
Keywords: tigecycline; complicated intra-abdominal infections (cIAI); complicated skin and soft tissue infections (cSSTI).
MeSH Terms: conditions — Intraabdominal Infections; Skin Diseases, Infectious; Soft Tissue Infections | interventions — Tigecycline

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients hospitalized because of cIAI or cSSTI
  Interventions: Drug: Tigecycline

INTERVENTIONS:
Drug: Tigecycline — Tigecycline 50 or 100 mg intravenously. Therapy conducted according to the package leaflet of Tygacil and to international treatment guidelines. Tygacil will be dosed according to labeling. The administration and duration of the therapy will be determined by the treating physician to meet the patient individual needs for treatment.
  Other Names: Tygacil

SUMMARY:
This is a study to evaluate the safety of tigecycline in patients with complicated intra-abdominal infections (cIAI) and complicated skin and soft tissue infections (cSSTI) under real practice in the usual hospital setting and patients' conditions, in order to assess the "real incidence" of adverse events related with tigecycline in these patients.

DETAILED DESCRIPTION:
Since around 50 patients were included in Spanish centers involved in the Phase III Tygacil clinical development program, and on the basis of the recruitment capacity of the centers within the predefined time window and the number of patients consenting to be enrolled in the study, the total number of patients estimated to be enrolled in the study is 500. With this sample size, it will be possible to obtain precise estimations of the incidence of particular types of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed by patients prior to this study entry.
* 18 years of age or older at the screening visit.
* Patients with cIAI or cSSTI.
* Patients who are going to or have just been given in the previous 48 hours at least a dose of tigecycline to treat any of the above infections.
* In the opinion of the investigator, the patient will be able to comply with the requirements of the protocol.

Exclusion Criteria:

* Known hypersensibility to tigecycline.
* Females who are pregnant, breast feeding, or at risk of pregnancy and not using a medically acceptable form of contraception.
* Use any investigational drug within four weeks of the screening visit.
* Uncooperative patients or a history of poor compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized because of complicated intra-abdominal infections (cIAI) or complicated skin and soft tissue infections (cSSTI), in the usual health care setting
Sampling Method: Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2008-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- [Derived] Bassetti M, Eckmann C, Bodmann KF, Dupont H, Heizmann WR, Montravers P, Guirao X, Capparella MR, Simoneau D, Sanchez Garcia M. Prescription behaviours for tigecycline in real-life clinical practice from five European observational studies. J Antimicrob Chemother. 2013 Jul;68 Suppl 2:ii5-14. doi: 10.1093/jac/dkt140. PMID 23772047
- [Derived] Guirao X, Sanchez Garcia M, Bassetti M, Bodmann KF, Dupont H, Montravers P, Heizmann WR, Capparella MR, Simoneau D, Eckmann C. Safety and tolerability of tigecycline for the treatment of complicated skin and soft-tissue and intra-abdominal infections: an analysis based on five European observational studies. J Antimicrob Chemother. 2013 Jul;68 Suppl 2:ii37-44. doi: 10.1093/jac/dkt143. PMID 23772045
- [Derived] Montravers P, Bassetti M, Dupont H, Eckmann C, Heizmann WR, Guirao X, Garcia MS, Capparella MR, Simoneau D, Bodmann KF. Efficacy of tigecycline for the treatment of complicated skin and soft-tissue infections in real-life clinical practice from five European observational studies. J Antimicrob Chemother. 2013 Jul;68 Suppl 2:ii15-24. doi: 10.1093/jac/dkt141. PMID 23772042
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1811048&StudyName=Post-Authorization%20Study%20Evaluating%20Safety%20Of%20Tigecycline

RESULTS

PARTICIPANT FLOW:
Groups:
- Complicated Skin and Soft-tissue Infections: Participants with Complicated Skin and Soft-tissue Infections (cSSTI) received tigecycline (Tygacil) at an initial dose of 100 milligram (mg) followed by 50 mg every 12 hours intravenously for 5 to 14 days based on local prescribing practices.
- Complicated Intra-Abdominal Infections: Participants with Complicated Intra-Abdominal Infections (cIAI) received tigecycline (Tygacil) at an initial dose of 100 mg followed by 50 mg every 12 hours intravenously for 5 to 14 days based on local prescribing practices.
Period: Overall Study
Arm/Group | Complicated Skin and Soft-tissue Infections | Complicated Intra-Abdominal Infections
Started | 19 | 96
Completed | 15 | 85
Not Completed | 4 | 11
Not completed — Exitus | 1 | 8
Not completed — Other | 1 | 3
Not completed — Pathogen not susceptible | 1 | 0
Not completed — Lack of effectiveness | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Complicated Skin and Soft-tissue Infections | Complicated Intra-Abdominal Infections | Total
Number analyzed (Participants) | 19 | 96 | 115
Age Continuous [Mean (Standard Deviation); unit: years] | 61.53 (11.01) | 59.27 (16.47) | 59.64 (15.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 47 | 52
  Male | 14 | 49 | 63

OUTCOME MEASURES:

1. Secondary Outcome: Percentage of Participants With Clinical Response of Cure
Description: Cure was defined as complete resolution of infection symptoms and clinical signs of the disease to the extent that no further antibiotic treatment was required, as assessed by the attending physician.
Time Frame: Days 2-5, 7-14 and 21-28 during treatment and Days 1-3 after end of treatment
Population: Intent-To-Treat (ITT) population included all evaluable participants who had at least one dose of study medication and one evaluation visit. 'n' signifies those participants who were evaluated for this measure at specified time points for each group respectively.
Measure: Number; unit: percentage of participants
Arm/Group | Complicated Skin and Soft-tissue Infections | Complicated Intra-Abdominal Infections
Number analyzed (Participants) | 19 | 96
percentage of participants
  On Days 2 to 5 (n= 19, 94) | 10.5 | 18.1
  On Days 7 to 14 (n= 13, 70) | 46.2 | 42.9
  On Days 21 to 28 (n= 6, 32) | 66.7 | 68.8
  On Days 1 to 3 after end of treatment (n= 19, 96) | 68.4 | 76.0

2. Secondary Outcome: Number of Participants With Susceptible Microbiological Pathogens
Description: Evaluation of susceptibility to the tigecycline treatment included: Escherichia coli Extended Spectrum Beta Lactamases (E. coli ESBL); Klebsiella pneumoniae (K. pneumoniae) ESBL; Bacteroides species resistant to clindamycin (RClin); Staphylococcus aureus (S. aureus) methicillin resistant S. aureus (MRSA); vancomycin resistant Enterococcus (VRE) species; Resistant to third generation cephalosporins (RCef3) Enterobacter species; RCef3 Serratia species; Proteus species ESBL; carbapenem resistant (RCarb) Pseudomonas aeruginosa (P. aeruginosa); Acinetobacter baumannii (A. baumannii) RCarb.
Time Frame: Baseline and Week 12
Population: Data was not summarized since the number of susceptibility tests to tigecycline during the study was extremely low.
Measure: Number; unit: participants
Arm/Group | Complicated Skin and Soft-tissue Infections | Complicated Intra-Abdominal Infections
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Any untoward medical occurrence in a participant who received study treatment was considered an AE without regard to possibility of causal relationship. An AE resulting in any of the following outcomes, or deemed to be significant for any other reason, was considered to be a SAE: death; initial or prolonged inpatient hospitalization; a life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Up to Week 12
Population: Safety population included all evaluable participants who received at least one dose of study medication and had at least one evaluation visit.
Measure: Number; unit: participants
Arm/Group | Complicated Skin and Soft-tissue Infections | Complicated Intra-Abdominal Infections
Number analyzed (Participants) | 19 | 96
participants
  AEs | 11 | 45
  SAEs | 4 | 28

4. Secondary Outcome: Number of Participants With Eradication of Microbiological Pathogens
Description: Evaluation of eradication after treatment with tigecycline included following microbiological pathogens: E. coli ESBL; K. pneumoniae ESBL; Bacteroides species RClin; S. aureus (MRSA); Enterococcus species (VRE); Enterobacter species RCef3; Serratia species RCef3; Proteus species ESBL; P. aeruginosa RCarb; A. baumannii RCarb.
Time Frame: Week 12
Population: Data was not analyzed since the number of samples obtained for culture was very low.
Measure: Number; unit: participants
Arm/Group | Complicated Skin and Soft-tissue Infections | Complicated Intra-Abdominal Infections
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Complicated Skin and Soft-tissue Infections | Complicated Intra-Abdominal Infections
Serious Adverse Events (participants affected / at risk) | 4/19 | 28/96
Other Adverse Events (participants affected / at risk) | 7/19 | 23/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Complicated Skin and Soft-tissue Infections (N=19) | Complicated Intra-Abdominal Infections (N=96)
Intestinal fistula (Gastrointestinal disorders) | 0 | 3
Multi-organ failure (General disorders) | 0 | 3
Pyrexia (General disorders) | 0 | 3
Sepsis (Infections and infestations) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Platelet count decreased (Investigations) | 0 | 2
Perianal abscess (Infections and infestations) | 2 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Failure to anastomose (Injury, poisoning and procedural complications) | 0 | 2
Abscess (Infections and infestations) | 0 | 2
Wound evisceration (Gastrointestinal disorders) | 0 | 1
Treatment failure (General disorders) | 1 | 0
Stupor (Nervous system disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Peritonitis (Gastrointestinal disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1
Ill-defined disorder (General disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
C-reactive protein (Investigations) | 0 | 1
Blood creatinine abnormal (Investigations) | 0 | 1
Biliary tract disorder (Hepatobiliary disorders) | 0 | 1
Azotaemia (Renal and urinary disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Aplasia (General disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Abdominal sepsis (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal abscess (Infections and infestations) | 0 | 1
Non specified (General disorders) | 1 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Complicated Skin and Soft-tissue Infections (N=19) | Complicated Intra-Abdominal Infections (N=96)
Abdominal pain (Gastrointestinal disorders) | 0 | 10
Pyrexia (General disorders) | 0 | 5
Renal failure (Renal and urinary disorders) | 1 | 4
Wound infection (Injury, poisoning and procedural complications) | 0 | 5
White blood cell count (Investigations) | 0 | 5
Intestinal fistula (Gastrointestinal disorders) | 0 | 1
C-reactive protein (Investigations) | 1 | 2
Body temperature increased (Investigations) | 0 | 4
White blood cell count increased (Investigations) | 0 | 3
Ill-defined disorder (General disorders) | 1 | 1
C-reactive protein increased (Investigations) | 0 | 3
Vomiting (Gastrointestinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Platelet count increased (Investigations) | 0 | 2
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Device related infection (General disorders) | 0 | 2
White blood cell analysis increased (Investigations) | 1 | 0
Transaminases abnormal (Investigations) | 1 | 0
Soft tissue infection (Infections and infestations) | 1 | 0
Retching (Gastrointestinal disorders) | 0 | 1
Postoperative wound infection (Injury, poisoning and procedural complications) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Phlebitis (Vascular disorders) | 0 | 1
Paronychia (Skin and subcutaneous tissue disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Neutrophil count increased (Investigations) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
Grand mal convulsion (Nervous system disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1
Escherichia infection (Infections and infestations) | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1
Blood amylase increased (Investigations) | 0 | 1
Biliary fistula (Hepatobiliary disorders) | 0 | 1
Bacterial infection (Infections and infestations) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.